CLINICAL TRIAL: NCT03514407
Title: An Open-Label Phase 1b Study of the Safety, Tolerability, and Preliminary Antitumor Activity of INCB059872 in Participants With Relapsed or Refractory Ewing Sarcoma
Brief Title: A Study of INCB059872 in Relapsed or Refractory Ewing Sarcoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic Business Decision
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB 59872-103; 2018-000062-11 (EudraCT Number)
Record Dates: First submitted 2018-04-20; First posted 2018-05-02 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Relapsed Ewing Sarcoma
Keywords: Relapsed Ewing sarcoma; bromodomain-containing protein (BRD) inhibitor; lysine demethylase 1 (LSD1) inhibitor
MeSH Terms: conditions — Sarcoma, Ewing | interventions — INCB059872

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- INCB059872 (Experimental): INCB059872
  Interventions: Drug: INCB059872

INTERVENTIONS:
Drug: INCB059872 — Part 1: Initial cohort of INCB059872 administered every other day (QOD) at the protocol-defined starting dose, with subsequent cohort dose escalation based on protocol-defined criteria. Part 2: Expansion with the recommended dose from Part 1.

SUMMARY:
The purpose of this study is to evaluate the safety and preliminary antitumor activity of INCB059872 in participants with Ewing sarcoma who are refractory or relapsed from prior standard therapy and not eligible for further standard systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of Ewing sarcoma and have progressed on or after standard therapies.
* Must not be a candidate for potentially curative therapy or standard-of-care approved therapy.
* Measurable disease by computed tomography or magnetic resonance imaging based on RECIST 1.1 as determined by site radiology.
* Eastern Cooperative Oncology Group performance status 0 to 2.
* Willingness to avoid pregnancy or fathering children.

Exclusion Criteria:

* Receipt of anticancer medications, anticancer therapies, or investigational drugs within protocol-defined intervals before the first administration of study drug.
* Must have recovered (≤ Grade 2 or at pretreatment baseline) from adverse events (AEs) from previously administered therapies except for stable chronic toxicities (≤ Grade 2) not expected to resolve.
* Untreated brain or central nervous system (CNS) metastases or brain/CNS metastases that have progressed.
* Prior radiotherapy within 2 weeks of study treatment. A 1-week washout period is permitted for palliative radiation to non-CNS disease with medical monitor approval.
* Laboratory values outside the protocol-defined range at screening.
* History or evidence of bleeding disorder or active clinically significant bleeding requiring medical intervention.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2020-06-25 (Actual); Study Completion 2020-06-25 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | Screening through 30 days after last dose of study treatment, up to approximately 6 months.
  Defined as any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of a drug in humans, whether or not considered drug-related.

SECONDARY OUTCOMES:
Objective response rate | Up to approximately 6 months.
  Defined as the percentage of participants who have a complete response or partial response as determined by investigator assessment of response per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Cmax of INCB059872 | Up to approximately 2 weeks.
  Defined as maximum observed plasma concentration.
tmax of INCB059872 | Up to approximately 2 weeks.
  Defined as time to maximum concentration.
t½ of INCB059872 | Up to approximately 2 weeks.
  Defined as apparent terminal-phase disposition half-life.
Cl/F of INCB059872 | Up to approximately 2 weeks.
  Defined as apparent oral dose clearance.

CONTACTS AND LOCATIONS:
Overall Officials: Fred Zheng, MD, Study Director — Incyte Corporation
Locations (11):
- United States (5):
  - UCLA Jonsson Comprehensive Cancer, Los Angeles, California
  - Mayo Clinic Jacksonville - PPDS, Jacksonville, Florida
  - Columbia University Medical Center, New York, New York
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
- Italy (3):
  - Istituto Ortopedico Rizzoli, Bologna
  - Policlinico Sant'orsola-Malpighi, Bologna
  - Ospedale Pediatrico Bambino Gesu IRCCS, Rome
- Spain (2):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clínico San Carlos, Madrid
- The Christie NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No